CLINICAL TRIAL: NCT02420522
Title: The Use of Repetitive Transcranial Magnetic Stimulation in the Treatment of Mild Cognitive Impairment Due to Brain Injury
Brief Title: Magnetic Brain Stimulation in the Treatment of Mild Cognitive Impairment
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Low recruitment rates and timeline viability analysis.
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: B2014:134
Record Dates: First submitted 2015-04-14; First posted 2015-04-20 (Estimated); Last update posted 2021-10-08 (Actual); Status verified 2021-09

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Active-first (Experimental): Participants randomly assigned to this arm will receive one week of active Repetitive Transcranial Magnetic Stimulation prior to one week of Sham Transcranial Magnetic Stimulation, separated by at least one week.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation; Device: Sham Transcranial Magnetic Stimulation
- Sham-first (Experimental): Participants randomly assigned to this arm will receive one week of Sham Transcranial Magnetic Stimulation prior to one week of active Repetitive Transcranial Magnetic Stimulation, separated by at least one week.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation; Device: Sham Transcranial Magnetic Stimulation
- Full-course Active (Active Comparator): Participants in this arm will receive three weeks (30 session, twice-daily) of active Repetitive Transcranial Magnetic Stimulation. This arm will not involve random assignment.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — A non-invasive method of brain stimulation.
Device: Sham Transcranial Magnetic Stimulation — A device designed to look, sound, and feel like a real magnetic stimulation coil without actually stimulating the brain.
  Arms: Active-first; Sham-first

SUMMARY:
This is a pilot study to test the efficacy of repetitive transcranial magnetic stimulation (rTMS) on cognitive improvement in individuals with mild cognitive impairment (MCI). The main objective of this study is to investigate the ability of rTMS to produce cognitive improvement in individuals with MCI. A secondary objective is to determine whether individuals with MCI following mild brain trauma respond differently to rTMS treatment compared to individuals with non-trauma related MCI.

Participants will undergo both active and sham (placebo) rTMS treatment. Cognitive and psychological assessments will be administered before and after each week of rTMS therapy, for both active and sham conditions. Cognitive testing will include verbal, semantic, logic, visual, conceptual, and memory tasks.

DETAILED DESCRIPTION:
This is an open-label pilot study to test the efficacy of repetitive transcranial magnetic stimulation (rTMS) on cognitive improvement in individuals with mild cognitive impairment (MCI). 16 patients with trauma-related MCI and 16 patients with non-trauma-related MCI will be recruited. All patients will undergo one week of active rTMS stimulation and one week of sham stimulation, separated by at least one week. Each treatment week will consist of five consecutive daily stimulation sessions. The order of active versus sham treatment sessions will be counterbalanced across subjects within each group (i.e., half of the subjects in each group will receive active stimulation first and half will receive sham first). Cognitive and psychological assessments will be administered before and after each week of rTMS therapy, for both active and sham conditions.

Additional participants (n=32; 16 without TBI) will be recruited who are receiving a full course (30 sessions) of active rTMS treatment (without a sham intervention). These participants will complete the same cognitive testing as the sham-crossover group at three time-points: pre-treatment, mid-treatment (after session 16), and post-treatment (after session 30).

ELIGIBILITY:
Inclusion Criteria:

* Adults presenting with mild cognitive impairment (trauma and non-trauma related)

Exclusion Criteria:

* History of a psychotic episode
* History of neurological illness
* Active alcohol or substance abuse
* History of seizure disorder
* Currently pregnant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2015-09; Primary Completion 2017-12 (Actual); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Cognitive changes | Three weeks
  Cognitive changes will be monitored through the administration of a number of pencil-and-paper and computer-based tasks that will be performed before and after each treatment week.

CONTACTS AND LOCATIONS:
Overall Officials: Mandana Modirrousta, MD PhD FRCPC, Principal Investigator — University of Manitoba
Locations (1):
- St Boniface Hospital, Winnipeg, Manitoba, Canada